CLINICAL TRIAL: NCT04231981
Title: A Multicenter, Open-Label, Single-Arm, Phase II Clinical Trial to Evaluate the Efficacy and Safety of INCMGA00012 in Advanced Penile Squamous Cell Carcinoma.
Brief Title: Efficacy of INCMGA00012 in Penile Squamous Cell Carcinoma (ORPHEUS)
Acronym: ORPHEUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP239; 2019-001172-11 (EudraCT Number)
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Penile Cancer
Keywords: Penile Cancer; Penile squamous cell carcinoma; Locally advanced penile cancer; Metastatic penile cancer; Unresectable locally advanced penile cancer; Unresectable penile cancer; PSqCC; PSCC; Penile Cancer stage IV
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Patients will receive INCMGA00012 500 mg by intravenous infusion on Day1 of each cycle.
  Interventions: Drug: Retifanlimab

INTERVENTIONS:
Drug: Retifanlimab — INCMGA00012 500 mg will be administered on Day1 of each cycle (once every four weeks), for up to 2 years.
  Other Names: INCMGA0012

SUMMARY:
This is a multicenter, open-label, single-arm, phase II clinical trial to evaluate the efficacy and safety of INCMGA00012 in Advanced Penile Squamous Cell Carcinoma

DETAILED DESCRIPTION:
Men age ≥ 18 years with locally advanced unresectable or metastatic PSqCC stage 4 (i.e. T4 or N3 or M1) that are presenting with radiologic progression of disease (PD) following or not standard treatment with chemotherapy.

After signing the ICF and confirmed eligibility, patients will receive INCMGA00012 500 mg by intravenous infusion on Day1 of each cycle, once every four weeks for up to 2 years.

Patients will receive treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected every 3 months (± 14 days) from the last dose of investigational product until the end of study (EoS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients have been informed about the nature of study, and have agreed to participate in the study, and signed the informed consent form (ICF) prior to participation in any study-related activities.
2. Male patients ≥ 18 years of age at the time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
4. Life expectancy ≥12 weeks.
5. Histologically-proven PSqCC.
6. Locally advanced unresectable or metastatic stage 4 PSqCC that is not amenable to resection with curative intent (T4 or N3 or M1).
7. Radiological evidence of locally advanced or metastatic disease.
8. Patients must have measurable disease or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v.)1.1 criteria.
9. Patients must agree to provide a tumor tissue sample from a metastatic site or the primary tumor at the time of study entry, with the exception of patients whom tumor biopsies cannot be obtained (e.g., inaccessible tumor or subject safety concern) that may submit an archived tumor specimen only upon agreement from the Sponsor. If feasible, patients will also be given the option of providing a tumor tissue sample at disease progression from metastasis or primary tumor (if tumor biopsies cannot be obtained for inaccessible lesion or subject safety concern).
10. Willingness and ability to provide blood samples (liquid biopsy) at the time of inclusion, after 2 cycles of study treatment (C3D1), and upon PD or study termination.
11. Adequate organ function:

    1. Hematological: White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 75.0 x109/L, and hemoglobin > 9.0 g/dL.
    2. Hepatic: Bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (< 3 x ULN in the case of Gilbert's disease); aspartate transaminase (AST), and alanine transaminase (ALT) ≤ 2.5 times × ULN (in the case of liver metastases ≤ 5 × ULN); Albumin > 2.5 mg/mL.
    3. Renal: Serum creatinine ≤ 1.5 x ULN; alternately measured or calculated creatinine clearance ≥30 mL/min with creatinine levels >1.5 × institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance).
    4. Coagulation: Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN and International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
12. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
13. Subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study treatment.
14. Patients that have received prior chemotherapy regimens or radiotherapy for locally recurrent and/or metastatic disease are not excluded but patients naïve of systemic treatment can also be included.
15. For pretreated patients, last dose of chemotherapy administered ≥ 28 days from study entry.

Exclusion criteria

1. Locally PSqCC candidate for curative treatment.
2. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
3. Known hypersensitivity to any of the excipients of INCMGA00012.
4. Receipt of anticancer therapy or participation in another interventional clinical study within 28 days before the first administration of study drug; 6 weeks for mitomycin C.
5. Radiotherapy within 14 days of first dose of study treatment with the following caveat: 28 days for pelvic radiotherapy.
6. Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of any grade of alopecia and anemia not requiring transfusion support). Endocrinopathy, if well-managed, is not exclusionary and should be discussed with Sponsor's medical monitor.
7. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 4 weeks of start of study drug, or patients who have not recovered from the side effects of any major surgery, or patients who may require major surgery during the study.
8. Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated (e.g., radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
9. Cardiovascular: patients that have any of the following within 6 months of randomization: severe/unstable angina, myocardial infarction, symptomatic pericarditis, symptomatic congestive heart failure (New York Heart Association functional classification III-IV), cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism, coronary/peripheral artery bypass graft, ongoing cardiac dysrhythmias of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0 grade ≥2, including, ventricular arrhythmias -except for benign premature ventricular contractions-, supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication, any conduction abnormality requiring a pacemaker or any cardiac arrhythmia not controlled with medication.
10. Metabolic: Uncontrolled hyper/hypothyroidism or diabetes mellitus type 1 (T1DM). Patients with hypothyroidism stable on hormone replacement will not be excluded from the trial. Patients with controlled T1DM on a stable insulin regimen may be eligible for this study.
11. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or immunosuppressive therapy within seven days prior to study treatment initiation.
12. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

    Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic steroid replacement therapy (≤ 10 mg prednisone daily) for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Prior allogenic stem cell or solid organ transplantation.
14. Has received a live vaccine within 28 days of the planned start of study drug. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live-attenuated vaccines and are not allowed.
15. Active/history of pneumonitis requiring treatment with steroids or active/history of interstitial lung disease.
16. Active uncontrolled infection at the time of screening.
17. Latent tuberculosis determined by a positive TST followed by confirmation by pulmonologists.
18. Participants who are known to be human immunodeficiency virus (HIV)-positive, unless all of the following criteria are met:

    1. CD4-positive count ≥ 300/μL;
    2. Undetectable viral load;
    3. Receiving highly active antiretroviral therapy.
19. Active hepatitis A virus (HAV) (positivity for HAV IgM antibody), hepatitis B virus (HBV) (patients with negative hepatitis B surface antigen [HBsAg] test and a positive antibody to HBsAg [anti-HBsAg] test at screening are eligible) or hepatitis C virus (HCV) (patients with a positive antibody to hepatitis C [anti-HCV] are eligible only if polymerase chain reaction [PCR] is negative for virus hepatitis C ribonucleic acid [RNA]).
20. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 3 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, or other noninvasive or indolent malignancy, or cancers from which the participant has been disease-free for >1 year, after treatment with curative intent.
21. Patients have any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro, Principal Investigator — ICO- Hospitalet
Locations (13):
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milano., Milan
  - IRCCS Ospedale San Raffaele, Milan
  - AUSL Reggio Emilia, Reggio Emilia
- Spain (10):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO-Hospitalet, L'Hospitalet de Llobregat
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital 12 de octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2020 and August 2021, a total of 18 male patients with locally advanced unresectable or metastatic PSqCC stage 4 (i.e. T4 or N3 or M1)presenting radiologic PD and/or chemotherapy were enrolled at 9 sites. Due there's only one arm, all the patients received INCMGA00012 until disease progression, death or discontinuation from the study.
Pre-assignment Details: Male patients ≥ 18 years of age. ECOG Performance Status ≤ 1. Life expectancy ≥12 weeks. Histologically-proven PSqCC. Locally advanced unresectable/metastatic stage 4 PSqCC that is not amenable to resection with curative intent (T4 or N3 or M1). - Radiological evidence of locally advanced or metastatic disease. - Adequate organ function.
Period: Overall Study
Arm/Group | Interventional Arm
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Death | 16
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Men age ≥ 18 years with locally advanced unresectable or metastatic PSqCC stage 4 (i.e., T4 or N3 or M1) that are presenting with radiologic progression of disease (PD) following or not standard treatment with chemotherapy.
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.5 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 5
  Spain | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The primary efficacy endpoint for the study is the ORR. The ORR is defined as the number of patients with CR and PR divided by the number of patients in the analysis set. Tumor response will be defined as best response based on local investigator's assessment according to RECIST criteria v.1.1.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Participants
  Yes | 3
  No | 15

2. Secondary Outcome: Efficacy Determined by Clinical Benefit Rate (CBR)
Description: CBR is defined as the number of patients with CR, partial response (PR) or stable disease (SD) (for at least 12 weeks) divided by the number of patients in the analysis set.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Participants
  Yes | 4
  No | 14

3. Secondary Outcome: Efficacy Determined by Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study treatment until the first documented PD based on RECIST v1.1. or death due to any cause, whichever occurs first based on local investigator's assessment according to RECIST criteria v1.1.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
months | 2 [1.6 to 3.3]

4. Secondary Outcome: Efficacy Determined by 6-months PFS
Description: 6-months PFS rate is defined as the proportion of patients who are alive and progression-free at 6 months from the date of first dose of study treatment based on iRECIST criteria.
Time Frame: Baseline up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Participants | 2

5. Secondary Outcome: Efficacy Determined by Duration of Response (DoR)
Description: DoR is defined as the time from first documented CR or PR until disease progression or death from any cause, based on local investigator's assessment according to RECIST criteria v1.1.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Median (Full Range); unit: months
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
months | 3.3 [1.8 to 8.5]

6. Secondary Outcome: Efficacy Determined by Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study treatment until death by any cause or the last date the patient was known to be alive.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Participants | 17

7. Secondary Outcome: Efficacy Determined by Maximum Tumor Shrinkage
Description: Maximum tumor shrinkage is defined as the percentage of tumor shrinkage from baseline (obtained from the sum of largest diameters of the target lesions), based on local investigator's assessment according to RECIST criteria v1.1.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
percentage of change from baseline | 15.9 (49.1)

8. Secondary Outcome: Safety Adverse Events (AEs)
Description: Number of patients with treatment-related AEs (Grade 3 and 4 AEs and serious adverse events [SAEs]) by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Time Frame: From baseline until disease progression or treatment discontinuation, up to 10.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 18
Participants
  Related AEs | 5
  Related SAEs | 0
  Related Grade 3 or 4 AEs | 1
  Safe patients from related AEs | 12

ADVERSE EVENTS:
Time Frame: From baseline until disease progression or treatment discontinuation, plus 28 days of follow-up after discontinuation (up to approximately 11.3 months)
Description: The investigator or investigator's team will report all protocol defined SAEs and ECIs to the Sponsor (MedSIR) no later than 24 hours of any site study team staff becoming aware of the event. The full details of the SAE and/or ECI should be collected and fully documented using theSAE form. Follow-up information will be sent along with the SAE form, if available on the day the event is reported or as soon as possible.
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 16/18
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=18)
Cellulitis (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Superinfection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=18)
Transaminases increased (Investigations) | 1 (2)
Fatigue (General disorders) | 4 (8)
Xerosis (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT04231981/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT04231981/SAP_001.pdf
  • Informed Consent Form (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT04231981/ICF_002.pdf